CLINICAL TRIAL: NCT06453096
Title: The Prevalence of Personality Disorders in Outpatient Forensic Mental Health in the Netherlands
Acronym: PREVPDFOROUT
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Barbera Van Reijswoud, principal investigator and phd-student, Vrije Universiteit Brussel
Other Study IDs: BvRVUBdeeloz2
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Personality Disorders
Keywords: forensic; prevalence; outpatient
MeSH Terms: conditions — Personality Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: prevalence of personality disorders — the prevalence of personality disorders will be investigated with a retrospective study

SUMMARY:
Personality disorders are associated with increased risk of violence and recidivism. Since information about the prevalence of personality disorders in outpatient forensic mental health care is scarce, the prevalence numbers in the Netherlands will be registered, in retrospective.

DETAILED DESCRIPTION:
Mentally disturbed people who commit or are at high risk of committing a crime, are treated in forensic psychiatry in the Netherlands. Treatment aims at preventing recidivism or lowering the risk of committing a crime by treating the psychiatric or psychological problems. Some people are committed in a hospital to receive this forensic psychiatric treatment, but a large group is treated in an outpatient forensic health (OFMH) facility.

All diagnoses and additional offences are treated in forensic psychiatry. Diagnoses are usually established through the DSM-5 and include, for example, psychotic disorders, substance-related disorder or sexual dysfunction. The offences are for instance, aggressive behavior, sexual violence, acquisition crimes or behavior problems like stalking.

In the Netherlands the Risk Need Responsivity (RNR) model is used in all kinds of forensic treatment and also in OFMH. Besides working on the most common risk factors like substance abuse or problematic circumstances at school or work, recognizing psychiatric diagnoses is important because this can be a risk factor in itself. Mental health problems can be seen both as a criminogenic need or as a responsivity factor.

Personality disorder (PD) is one of the diagnoses that is important to recognize. PDs are associated with increased risk of violent and antisocial behavior, and with recidivism risk. PD's also require a specific treatment approach; therefore, there are programs that focus on this group. Knowledge about prevalence is important for several reasons. Prevalence studies show the disease burden of certain conditions and promote both the recognition of these and the formulation of policy in healthcare. Knowledge of prevalence rates can also help therapists to be more attentive to certain problems or diagnoses, such as PDs. Consequently, this knowledge can facilitate the identification of PDs, which also ensures that treatment approaches are better tailored to PDs. A systematic review of studies on detainees found that 46% of the men and 21 % of the women were diagnose with antisocial PD and 65% of the men and 42% of the women exhibited a PD, including antisocial PD. In forensic inpatients almost 78%* of the population had a PD with 28% a cluster B PD and 42% a PD not otherwise specified. So, prevalence figures in forensic populations are quite high. The question however arises whether PDs are also common among forensic outpatients in the Netherlands? Figures on prevalence of PDs in OFMH are however scarce. Therefore, this research aims at identifying the prevalence of PDs in OFMH in the Netherlands.

research question: What DSM-5 classifications have been made (primary and secondary)? How can the group with a PS be described with respect to gender, age, education, nationality, legal title, nature of offense and care received.

ELIGIBILITY:
Inclusion Criteria: information of all patients from forensic outpatients facilities who received care in 2023 in the Netherlands -

Exclusion Criteria: no

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients from forensic outpatients facilities who received care in 2023 in the Netherlands
Sampling Method: Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-23 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
prevalence of Personality disorders (PDs) | 2023
  PDs according to DSM 5 criteria in number of people and percentages

SECONDARY OUTCOMES:
socio demographic correlates | 2023
  gender, age, education, nationality in number of people and percentages
crime and sort of treatment | 2023
  indexcrime and form of treatment (For-fact or ambulatory) in number of people and percentages

CONTACTS AND LOCATIONS:
Overall Officials: Barbera van reijswoud, drs, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- VUB, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. (2022). Diagnostic and Statistical Manual of Mental Disorders (5th ed., text rev.). Author.
- [Background] Andrews, D. A., Bonta, J., & Wormith, J. S. (2011). The risk-need-responsivity (RNR) model: Does adding the good lives model contribute to effective crime prevention? Criminal Justice and Behavior, 38(7), 735-755. https://doi.org/10.1177/0093854811406356
- [Background] Borges Migliavaca C, Stein C, Colpani V, Barker TH, Munn Z, Falavigna M; Prevalence Estimates Reviews - Systematic Review Methodology Group (PERSyst). How are systematic reviews of prevalence conducted? A methodological study. BMC Med Res Methodol. 2020 Apr 26;20(1):96. doi: 10.1186/s12874-020-00975-3. PMID 32336279
- [Background] DJI. (2024). Overzicht door DJI gecontracteerde aanbieders FZ per 1/1/2024 per zorgsoort. https://www.forensischezorg.nl/documenten/publicaties/2024/02/12/overzicht-aanbieders-fz-2024-per-zorgsoort
- [Background] Douglas, K. S., Hart, S. D., Webster, C. D., Belfrage, H., Guy, L. S., & Wilson, C. M. (2014). Historical-Clinical-Risk Management-20, Version 3 (HCR-20V3): Development and Overview. International Journal of Forensic Mental Health, 13, 93-108. https://doi.org/DOI: 10.1080/14999013.2014.906519
- [Background] Drieschner, K., & Tollenaar, N. (2011). Recidive tijdens forensische zorgtrajecten 2013-2017. Cahier 2021-18. www.wodc.nl
- [Background] Fazel S, Danesh J. Serious mental disorder in 23000 prisoners: a systematic review of 62 surveys. Lancet. 2002 Feb 16;359(9306):545-50. doi: 10.1016/S0140-6736(02)07740-1. PMID 11867106
- [Background] Guyton, M. R., & Foerschner, A. (2017). Treatment of Personality Disorders in Forensic/Correctional Settings. In R. Roesch & A. N. Cook (Eds.), Handbook of Forensic Mental Health Services (pp. 290-322). Routledge. https://doi.org/10.4324/9781315627823-11
- [Background] ILOSTAT. (2011). ISCED. International Standard Classification of Education. https://ilostat.ilo.org/resources/concepts-and-definitions/classification-education/
- [Background] Jankovic M, Masthoff E, Spreen M, de Looff P, Bogaerts S. A Latent Class Analysis of Forensic Psychiatric Patients in Relation to Risk and Protective Factors. Front Psychol. 2021 Jul 20;12:695354. doi: 10.3389/fpsyg.2021.695354. eCollection 2021. PMID 34354640
- [Background] Lutz M, Zani D, Fritz M, Dudeck M, Franke I. A review and comparative analysis of the risk-needs-responsivity, good lives, and recovery models in forensic psychiatric treatment. Front Psychiatry. 2022 Oct 31;13:988905. doi: 10.3389/fpsyt.2022.988905. eCollection 2022. PMID 36386990
- [Background] Noland E, Strandh M. Historical, clinical and situational risk factors for post-discharge recidivism in forensic psychiatric patients - A Swedish registry study. Int J Law Psychiatry. 2021 Nov-Dec;79:101749. doi: 10.1016/j.ijlp.2021.101749. Epub 2021 Nov 10. PMID 34768026
- [Background] Tamam L, Ozpoyraz N, Karatas G. Personality disorder comorbidity among patients with bipolar I disorder in remission. Acta Neuropsychiatr. 2004 Jun;16(3):175-80. doi: 10.1111/j.1601-5215.2004.00074.x. PMID 26984171
- [Background] Taylor, J. (2014). Developing a framework for the identification of criminogenic needs in offenders with intellectual disability and personality disorder: The Treatment Need Matrix. Advances in Mental Health and Intellectual Disabilities, 8(1), 43-50. https://doi.org/10.1108/AMHID-07-2013-0051
- [Background] van den Bosch LM, Hysaj M, Jacobs P. DBT in an outpatient forensic setting. Int J Law Psychiatry. 2012 Jul-Aug;35(4):311-6. doi: 10.1016/j.ijlp.2012.04.009. Epub 2012 May 5. PMID 22560672
- [Background] Verschuur, J., & Keulen-de Vos, M. (2018). Basis zorgprogramma voor de forensische ambulante zorg.
- [Background] Yu R, Geddes JR, Fazel S. Personality disorders, violence, and antisocial behavior: a systematic review and meta-regression analysis. J Pers Disord. 2012 Oct;26(5):775-92. doi: 10.1521/pedi.2012.26.5.775. PMID 23013345
- [Background] Zimmerman M, Galione JN, Chelminski I, Young D, Dalrymple K, Morgan TA. Does the diagnosis of multiple Axis II disorders have clinical significance? Ann Clin Psychiatry. 2012 Aug;24(3):195-201. PMID 22860239
- [Background] Zorginstituut Nederland. (2022). Kwaliteitskader Forensische Zorg 2022-2028. https://www.rijksoverheid.nl/documenten/rapporten/2020/11/02/tk-bijlage-visie-forensische-zorg-2020.